CLINICAL TRIAL: NCT01384422
Title: Safety and Preliminary Efficacy of GLPG0634 in Methotrexate-refractory Active Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-201
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: methotrexate-refractory
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG0634 100 mg bid oral capsules (Experimental)
  Interventions: Drug: GLPG0634
- GLPG0634 200 mg qd oral capsules (Experimental)
  Interventions: Drug: GLPG0634
- Placebo oral capsules (Placebo Comparator)
  Interventions: Drug: GLPG0634

INTERVENTIONS:
Drug: GLPG0634

SUMMARY:
* Thirty six patients suffering from active rheumatoid arthritis despite continued treatment with methotrexate will be evaluated for improvement of disease activity when taking GLPG0634 or matching placebo for 4 weeks.
* During the course of the study, patients will also be examined for any side effects that may occur, and the amount of GLPG0634 present in the blood as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Have active RA as shown by five or more swollen joints (from the 66-joint count), five or more tender joints (from 68-joint count), and a serum CRP ≥1.0 mg/dL;
* Have received methotrexate for six months or longer and at a stable dose of 7.5 to 25 mg/week (extremes included) for at least four weeks prior to screening and willing to continue on this regimen for the duration of the study;
* If taking oral steroids, these should be at a dose ≤10 mg/day of prednisone or prednisone equivalent and stable for at least four weeks prior to screening;
* If taking non-steroidal anti-inflammatory drugs (NSAIDs), these must be at a stable dose for at least two weeks prior to screening;
* Female subjects must have a negative pregnancy test unless they are surgically sterile or have been post-menopausal for at least one year (12 consecutive months without menses);
* Women of childbearing potential must use a medically acceptable means of birth control and agree to continue its use during the study and for at least four weeks after the last dose of study drug. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue its use for at least 3 months after the last dose of study drug; and
* Able and willing to sign the informed consent prior to screening evaluations and agree to schedule of assessments.

Exclusion Criteria:

* Treatment with disease-modifying antirheumatic drugs (DMARDs), other than background methotrexate;
* Current or previous RA treatment with a biological agent, with the exception of biologics administered in a clinical study setting more than six months prior to screening (12 months for rituximab or other B cell depleting agents);
* Previous treatment at any time with a cytotoxic agent, other than methotrexate, before screening;
* Receipt of an intra-articular or parenteral corticosteroid injection within four weeks prior to screening;
* Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the Investigator, such as anaphylaxis, requiring hospitalization;
* Positive serology for human immunodeficiency virus (HIV)1 or 2 or hepatitis B or C, or any history of hepatitis from any cause with the exception of hepatitis A;
* History of any inflammatory rheumatological disorders other than RA;
* History of tuberculosis (TB) infection;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The number of patients with an ACR20 score at Week 4 as a measure of efficacy | 4 weeks
  To preliminarily evaluate the efficacy of GLPG0634 compared to placebo in terms of the proportion of subjects achieving an ACR20 response at Week 4

SECONDARY OUTCOMES:
The number of patients with ACR20/50/70 response, time to response and DAS28 score at every visit as a measure of efficacy
  To evaluate the efficacy of GLPG0634 compared to placebo in terms of ACR response criteria at every visit (ACR20, ACR50, ACR70), time to response, and disease status (DAS28[C-reactive protein, CRP]
The number of patients with adverse events, abnormal lab tests, vital signs and ECG as a measure of safety and tolerability
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms of adverse events (AEs), laboratory test abnormalities, vital signs and electrocardiogram (ECG)
The plasma levels of GLPG0634 as a measure of PK and the levels of immune- and inflammation-related parameters in blood as a measure of PD
  To characterize the pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0634 in subjects with rheumatoid arthritis (RA)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV
Locations (1):
- Innophar MO S.R.L., Chisinau, Moldova

REFERENCES:
- [Derived] Vanhoutte F, Mazur M, Voloshyn O, Stanislavchuk M, Van der Aa A, Namour F, Galien R, Meuleners L, van 't Klooster G. Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Filgotinib, a Selective JAK-1 Inhibitor, After Short-Term Treatment of Rheumatoid Arthritis: Results of Two Randomized Phase IIa Trials. Arthritis Rheumatol. 2017 Oct;69(10):1949-1959. doi: 10.1002/art.40186. Epub 2017 Aug 31. PMID 28622463
- [Derived] Namour F, Diderichsen PM, Cox E, Vayssiere B, Van der Aa A, Tasset C, Van't Klooster G. Pharmacokinetics and Pharmacokinetic/Pharmacodynamic Modeling of Filgotinib (GLPG0634), a Selective JAK1 Inhibitor, in Support of Phase IIB Dose Selection. Clin Pharmacokinet. 2015 Aug;54(8):859-74. doi: 10.1007/s40262-015-0240-z. PMID 25681059